CLINICAL TRIAL: NCT00865397
Title: Observational Study of Glycaemic Control in Type 2 Diabetic Patients Uncontrolled on Oral Antidiabetic Agents and Starting With Once Daily Levemir® (Insulin Detemir) - 24 Weeks, Prospective, Multicentre Observational Study in Hungary
Brief Title: Observational Study in Type 2 Diabetics Failing on Oral Antidiabetic Therapy and Starting on Insulin Treatment
Acronym: HA-BOT
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN304-3699
Record Dates: First submitted 2009-03-18; First posted 2009-03-19 (Estimated); Last update posted 2016-11-23 (Estimated); Status verified 2016-11

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Insulin Detemir

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A
  Interventions: Drug: insulin detemir

INTERVENTIONS:
Drug: insulin detemir — Effectiveness data collection in connection with the use of the drug Levemir® in daily clinical practice.
  Other Names: Levemir®; NN304

SUMMARY:
This study is conducted in Europe. The aim of this observational study is to evaluate glycaemic control in subjects with type 2 diabetes using once daily Levemir® as initiation of insulin therapy in Hungary.

ELIGIBILITY:
Inclusion Criteria:

* Patient with type 2 diabetes inadequately controlled by OAD therapy based on the discretion of individual physician
* Patient willing to sign informed consent
* Particular attention should be paid to age limits, indications and contraindications and the drug interactions that are listed within the product labels

Exclusion Criteria:

* Subjects with diagnosed type 1 diabetes mellitus
* Subjects who are unlikely to comply with observational plan, (e.g., uncooperative attitude, inability to return for further visits)
* Subjects with hypersensitivity to Levemir® or to any of the ingredients
* Women of childbearing potential, who are pregnant, breast-feeding or intend to become pregnant within next 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A non-randomised sample of approximately 1000 subjects with OAD failure from specialists - diabetologists practice who have been deemed appropriate to receive insulin detemir as add-on to OAD therapy as part of routine out-patient care by the prescribing physician.
Sampling Method: Non-Probability Sample
Enrollment: 1032 (Actual)
Dates: Start 2009-02; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c | after 24 weeks

SECONDARY OUTCOMES:
Percentage of subjects to reach HbA1c below 7.0% and equal to or more than 6.5% | after 12 weeks and 24 weeks
Change in FPG (Fasting Plasma Glucose) | after 12 weeks and 24 weeks
Change in body weight | after 12 weeks and 24 weeks
Change in waist and hip circumference | after 12 weeks and 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Budapest, Hungary

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com